CLINICAL TRIAL: NCT03526718
Title: Improved Understanding of Ongoing Transmission of Leprosy in the Comoros, a Region Hyperendemic for the Disease.
Brief Title: Improved Understanding of Ongoing Transmission of Leprosy in the Hyperendemic Comoros (ComLep)
Acronym: ComLep
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Damien Foundation (Other); Programme National de lutte contre la Lèpre et la Tuberculose, Comores (Unknown); Instituto Oswaldo Cruz (Unknown); R2STOP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1147/16
Record Dates: First submitted 2018-04-23; First posted 2018-05-16 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Leprosy
Keywords: Transmission; Genotyping; Risk factors
MeSH Terms: conditions — Leprosy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Skin biopsy (non facial), Nasal swabs, Fingerstick blood and Slit skin smears (non facial and only for multibacillary patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite decades of a solid leprosy control program, including active case finding and follow-up on therapeutic outcome, the Comoros islands of Anjouan and Moheli continue to be hyperendemic for leprosy, with leprosy case notifications far exceeding those for tuberculosis, while the third island, Grande Comore, presents few cases. The high proportion (31% in 2015) of disease in children indicates that recent transmission is a major driver of the persistent endemicity, and that present control measures are not sufficient. The low proportion (2.6% average in last 10 years) of grade II disabilities in newly diagnosed cases indicates that case detection is early.

The main objective of the present proposal is to identify which persons would most benefit from prophylactic treatment. The secondary objective is to unravel human, bacterial and environmental risk factors for transmission of and progression to leprosy disease, with the ultimate goal to reduce the leprosy incidence.. The program has remaining expertise to re-establish laboratory confirmation of leprosy patients, allowing to optimize and validate molecular genotyping techniques to complement conventional epidemiological investigations in a 3-year prospective cohort of leprosy patients and their close contacts, aiming to identify transmission links. A third objective is to document diagnostic delays in more detail

As the leprosy control programme has initiated a pilot study on rifampicin prophylaxis in four villages on Anjouan in 2015, a prospective cohort study will permit measuring the leprosy incidence in close contacts as well as those in neighboring houses, who did or did not receive rifampicin prophylaxis.

The expected outcome of this project will be to identify risk factors for leprosy transmission. Specifically, we expect to identify those contacts at highest risk of developing leprosy disease, who would most benefit from rifampicin prophylaxis or other preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* in the prospective cohort study: All newly diagnosed leprosy patients (any age) on the island of Anjouan who provide written informed consent.
* In the in-depth interviews: Patients who are part of a cluster and provide written informed consent. Additional written informed consent will be asked for questions in which the identity of other member(s) of a cluster needs to be revealed.

Exclusion Criteria:

* in the prospective cohort study: None.
* In the in-depth interviews: Patients belonging to clusters not extending beyond the same first or second circle

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Comoros islands, located between Madagascar and Mozambique, continue to be hyperendemic for leprosy. Periodic active case finding across the entire island of Anjouan is in place, resulting in early case detection, and every patient identified is being treated with highly effective multi drug therapy. Nevertheless, the high proportion of leprosy in children (31% were <15y old in 2015) in combination with a low relapse rate (<2%) indicate transmission continues unabated. The majority of the patients in Anjouan are paucibacillary.
Sampling Method: Probability Sample
Enrollment: 889 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Leprosy incidence among contacts of an index patient | The incidence rate ratio will be recorded during the 3-year recruitment period op the study.
  Incidence rate ratios among the contacts by proximity to the index patients will be calculated. Classification of contacts in proximity groups is a dynamic process. Persons belonging to the same household, surrounding households, entire village, or entire island may shift to closer proximity groups when leprosy patients are diagnosed in their environment. Since date of diagnosis, and any recent migration, will be recorded for each patient, we will be able to reallocate contacts to other circles and attribute to each contact a period of exposure within each circle.

SECONDARY OUTCOMES:
Recent transmission cluster | All the samples over the three years should be analysed the able to fully explore the transmission links. Therefore, this outcome will be assessed through study completion, which will probably take1 year.
  Transmission links will be defined as identical genotypes based on their "variable number of tandem repeat(VNTR)"- profile. The definition of clustering will be based on comparison of the copy number of the VNTRs using two different stringencies: either considering those that presented identical copy number for all 17 alleles, or considering those that had identical copy number excluding the most variable loci.
Patient and health system delay. | This outcome can be calculated at the end of the recruitment phase of the study.Therefore, this outcome will be assessed through study completion, which will probably take1 year.
  Mean patient and health systems delay with 95% confidence interval will be calculated. The questionnaire will comprise questions on the duration of the symptoms and the health seeking behavior of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Bouke C de Jong, MD,PhD, Principal Investigator — Institute of Tropical Medicine
Locations (1):
- Damien Foundation, Moutsamoudou, Ndzuwani, Comoros

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be considered once the datasets are locked at time of publication.

REFERENCES:
- [Derived] Marijke Braet S, Jouet A, Aubry A, Van Dyck-Lippens M, Lenoir E, Assoumani Y, Baco A, Mzembaba A, Cambau E, Vasconcellos SEG, Rigouts L, Suffys PN, Hasker E, Supply P, de Jong BC. Investigating drug resistance of Mycobacterium leprae in the Comoros: an observational deep-sequencing study. Lancet Microbe. 2022 Sep;3(9):e693-e700. doi: 10.1016/S2666-5247(22)00117-3. Epub 2022 Jul 15. PMID 35850123